CLINICAL TRIAL: NCT05872087
Title: Comparative Study Between Nebulised Dexmedetomidine and Nebulised Midazolam in Reducing Preoperative Anxiety and Emergence Delirium in Children Undergoing Lower Abdominal Surgeries
Brief Title: Comparative Study Between Nebulised Dexmedetomidine and Nebulised Midazolam in Children Undergoing Lower Abdominal Surgeries
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: midazolam vs dexmedetomidine
Record Dates: First submitted 2023-03-22; First posted 2023-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2023-05

CONDITIONS: Emergence Delirium; Anxiety Preoperative
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine (Active Comparator): will receive nebulized Dexmedetomidine 3 µg/kg
  Interventions: Drug: Nebulised Dexmeditomidine
- Midazolam (Active Comparator): will receive nebulized Midazolam 0.3 mg/kg
  Interventions: Drug: Nebulised Midazolam

INTERVENTIONS:
Drug: Nebulised Dexmeditomidine — premedication by dexmeditomidine 3mcg/kg in children undergoing lower abdominal surgeries
  Other Names: premedication by nebulised dexmeditomidine
  Arms: Dexmedetomidine
Drug: Nebulised Midazolam — premedication by nebulised midazolam 0.3mg/kg in children undergoing lower abdominal surgeries
  Other Names: Premedication by nebulised midazolam
  Arms: Midazolam

SUMMARY:
Comparative study between nebulised dexmedetomidine and nebulized midazolam in reducing preoperative anxiety and emergence delirium in children undergoing lower abdominal surgeries

DETAILED DESCRIPTION:
Dexmedetomidine is widely used in children and is replacing midazolam as the drug of choice for preoperative anxiolysis and sedation. However, there are limited studies comparing nebulized route in reducing preoperative anxiety and emergence delirium in children undergoing lower abdominal surgeries

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3-8 years
* ASA I&II
* Undergoing lower abdominal surgeries for example hernia repair and circumcision

Exclusion Criteria:

* Children with chest infection, respiratory disease, cardiac disease
* Children with mental or physical disabilities, treatment with sedatives and anticonvulsants
* Parental refusal
* Allergy to study drugs

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
level of preoperative anxiety | 30 minutes after drug administration
  The level of anxiety of the child during separation from parents according to Parental separation anxiety scale (PSAS), with a 4-point scale as: 1=easy separation; 2=whimpers, but is easily reassured, not clinging; 3=cries and cannot be easily reassured, but not clinging to parents and 4=crying and clinging to parents
Incidence of emergence delirium | immediate postoperative
  Incidence of emergence delirium, wake up behaviour will be assessed according to Watcha scale where Score is observed values as follows: 0= asleep, 1=calm, 2=crying but can be consoled, 3=crying but cannot be consoled, 4=agitating and thrashing around

SECONDARY OUTCOMES:
the level of sedation | 30 minutes after drug administration
  The level of sedation when the child first seen in the operating room 30 minutes after sedation using Ramsey sedation scale
hemodynamic changes | perioperative
  number of participants experienced any hemodynamic changes if more than 20% change in mean arterial pressure (MAP) and Heart Rate (HR).
PONV | perioperative
  Incidence of post-operative nausea and vomiting.
recovery time | up to 2 hours postoperative
  Recovery time, time between laryngeal mask removal and discharge from recovery room.
total fentanyl use | intraoperative
  Total fentanyl use during operation

CONTACTS AND LOCATIONS:
Locations (1):
- Ainshams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No